CLINICAL TRIAL: NCT00739479
Title: CCRC: Effects of Partially Hydrolyzed Whey Peptides (PHWP) On Weight Loss In Individuals With The Metabolic Syndrome (METS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidika E. Karakas, MD (Other)
Collaborators: California Dairy Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Sidika E. Karakas, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200816190-1
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2008-08

CONDITIONS: Metabolic Syndrome; Overweight
Keywords: Metabolic Syndrome; METS; Obesity; Partially Hydrolyzed Whey Protein; Partially Hydrolyzed Gelatin; PHWP; PHG; Weight Loss
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients will be randomized to receive PHWP. Since sex and baseline weight can influence the response, randomization will be stratified according to these variables.
  Interventions: Dietary Supplement: Weight Loss
- 2 (Placebo Comparator): Patients will be randomized to receive PHG. Since sex and baseline weight can influence the response, randomization will be stratified according to these variables.
  Interventions: Dietary Supplement: Weight Loss

INTERVENTIONS:
Dietary Supplement: Weight Loss — Participants will reduce their total dietary intake by ~800 kcal/day. ~100 kcal will be replaced by either the PHWP of PHG protein supplement, resulting in a total energy restriction of ~700 kcal/day.

SUMMARY:
The aim of this study is to compare the effects of two different protein supplements (partially hydrolyzed whey protein, PHWP vs. partially hydrolyzed gelatin, PHG) on weight loss in obse individuals with metabolic syndrome (METS). These two supplements will contain equal amounts of protein but differ considerably in their amino acid contents. Whey protein is rich in essential amino acids whereas gelatin is rich in proline.

In obese individuals with METS, the hypotheses are:

* PHWP will augment fat-mass loss and increase lean-mass to fat-mass ration more than PHG.
* PHWP will improve insulin action more than PHG.
* PHWP will decrease cardiovascular disease risk more than PHG.

DETAILED DESCRIPTION:
The Metabolic Syndrome (METS) is a clinical disorder characterized by the following problems: Obesity, especially located in the waist area, elevated blood fats (lipids), high blood pressure and insulin resistance. The METS affects one third of the adult population in the USA and increases the risks for both diabetes and hardening of the arteries, leading to heart attacks and strokes.

The best treatment for improving the symptoms of METS is weight loss. In previous studies, it has been demonstrated that whey protein (WP) supplementation increased weight loss and especially fat-mass loss in obese, insulin resistant women when compared to carbohydrates. We now propose to compare WP to another protein source in patients with the METS during weight loss. In addition, we will use a special preparation called partially hydrolyzed whey protein, which may have specific properties that increase fat mass loss.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnoses of Metabolic Syndrome (at least 3/5 of the following)

  * Waist Circumference: men: >40 in women: >35 in
  * Blood Pressure: >135/>85 mm Hg
  * Triglycerides: >150 mg/dl
  * HDL-cholesterol: men: <40 mg/dl women: <50 mg/dl
  * Fasting Glucose: >100 mg/dl
* Ages 18 to 65 Years
* BMI range of 27 to 42 kg/m^2
* Body weight <300 lbs
* Weight Stable for 3 Months

Exclusion Criteria:

* Subjects who habitually consume protein supplements or have eating disorders
* Recent delivery (within 12 months), lactation, pregnancy or intention to become pregnant
* Type 2 diabetes, kidney disease, liver disease, anemia, gout, cancer, untreated thyroid disease, gastrointestinal disease, other metabolic diseases or malabsorption syndromes
* Triglyceride >500 mg/dl, Cholesterol >260 mg/dl
* Use of insulin sensitizers, lipid lowering medication or ACE inhibitors
* Use of anti-obesity medications or supplements for at lease 6 months prior to start of study
* Known allergy or adverse reaction to protein and dairy products (including lactose)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The investigators hope to determine the effects of incorporating PHWP into the diet of a person diagnosed with METS. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Sidika E Kasim-Karakas, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis CCRC, Sacramento, California, United States

REFERENCES:
- [Derived] Piccolo BD, Comerford KB, Karakas SE, Knotts TA, Fiehn O, Adams SH. Whey protein supplementation does not alter plasma branched-chained amino acid profiles but results in unique metabolomics patterns in obese women enrolled in an 8-week weight loss trial. J Nutr. 2015 Apr;145(4):691-700. doi: 10.3945/jn.114.203943. Epub 2015 Feb 4. PMID 25833773
- [Derived] Comerford KB, Buchan W, Karakas SE. The effects of weight loss on FABP4 and RBP4 in obese women with metabolic syndrome. Horm Metab Res. 2014 Mar;46(3):224-31. doi: 10.1055/s-0033-1353204. Epub 2013 Aug 26. PMID 23979787
- See also: UC Davis Website - Featured Clinical Trials — http://www.ucdmc.ucdavis.edu/clinicaltrials/